CLINICAL TRIAL: NCT02205684
Title: Effects of Aerobic High Intensity Training on Symptoms, Cognition, Cortical Structure, Substance Use and Metabolic Indices in Patients With Schizophrenia Spectrum Disorder
Brief Title: Effects of Physical Activity in Psychosis
Acronym: EPHAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); Norwegian Research network in Severe Mental Illness (Unknown)
Responsible Party: Principal Investigator, John Abel Engh, Principal Investigator, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/372/REK sør-øst C
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Substance Use
Keywords: Physical activity; Exercise; High intensity training; Schizophrenia; Symptoms; Well-being; Cognition; Hippocampal volume; Neuroplasticity; Smoking; Substance use; Metabolic indices
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders; Motor Activity; Smoking | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity (Experimental): Aerobic High Intensity Training (HIT)
  Interventions: Other: Physical activity
- Computer game skills training (Active Comparator): Playing Nintendo Wii Sports
  Interventions: Other: Computer game skills training

INTERVENTIONS:
Other: Computer game skills training — Playing Nintendo Wii Sports
  Arms: Computer game skills training
Other: Physical activity — Aerobic High Intensity Training (HIT)
  Arms: Physical activity

SUMMARY:
Physical health problems are common in schizophrenia with a two- to three-fold increased morbidity and mortality rate, resulting in a 20 years reduction in life expectancy. A genetic vulnerability for developing cardiovascular disease has been documented in these patients, and many lifestyle factors also negatively influence physical health. Patients with schizophrenia are likely to smoke, are physically inactive and overweight, suffer from malnutrition due to unhealthy diet, and have reduced cardiorespiratory fitness. Moreover, these patients have increased risk of developing diabetes mellitus type II and metabolic syndrome. These aspects demonstrate the need for multi-disciplinary treatments of patients with schizophrenia and underline the need for addressing their physical health.

Poor physical fitness seems to be associated with exacerbated negative symptoms and increased cognitive dysfunction in patients with schizophrenia. However, evidence on physical activity and its consequences in schizophrenia is scarce. In this randomized controlled trial we investigate the effects of high intensity training in outpatients with schizophrenia on psychotic symptoms and well-being, cognition and cortical structure, tobacco smoking and substance use, in addition to metabolic indices.

DETAILED DESCRIPTION:
Outpatients in treatment will be recruited in this randomized controlled trial (RCT). The patients will be randomized to either a Computer gaming Skills Group (CSG) or to a physical Exercise Group (EG). The groups are identically organized in two locations. The interventions last for 12 weeks, and treatment as usual will be continued for all patients. Patients will be assessed when entering the study (after randomization and allocation to one of the clinical groups), as well as post-treatment and 4 months post-treatment. Thus, the planned study is prospective with a longitudinal design. It is single blind in the sense that the assessment of psychiatric symptom level and neurocognitive function will be performed by research staff blind for group membership. The physiological testing will be performed by staff involved in training and will not be blinded.

EG participants will perform aerobic high intensity training (HIT) consisting of supervised walking/running on a treadmill 2 times a week for 12 weeks. Each session will have the following structure; eight-minute warm-up, followed by four times four minutes intervals with 85-95% of maximum heart rate, with active pauses of three minutes of walking at 70% of maximum heart rate. The exercise session will end with a five minute cool-down period. HIT performed as 4 x 4 intervals has been proven feasible and safe among patients with schizophrenia and in other clinical populations.

Participants in the CSG take part in sessions in the clinic playing computer games (Nintendo Wii Sports). The time spent with activities in the clinic will be the same in both groups. When absent from scheduled physical exercise/playing computer games the subjects will be offered to participate on a following day. If absent for a whole week, the training period/computer games playing period will be prolonged accordingly.

In this randomized controlled trial we investigate the effects of HIT in outpatients with schizophrenia on symptoms and well-being, cognition and brain structure, smoking habits and substance use, as well as metabolic indices.

The participating outpatient clinics are catchment area based and cover a population of 200 000 persons with more than 250 patients in the diagnostic group in treatment at one time.

ELIGIBILITY:
Inclusion Criteria:

* verified (Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, SCID) diagnosis of schizophrenia spectrum disorder
* outpatient in treatment
* written informed consent
* fluent in a Scandinavian language

Exclusion Criteria:

* chest pain during exercise
* unstable angina pectoris
* suspicion of recent myocardial infarction
* uncontrollable arrhythmia
* acute infection with lymphadenopathy
* malignant hypertension
* neurological disorder
* severe physical disability
* medical condition incompatible with particiption
* comorbid diagnosis of mild mental retardation
* pregnancy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Cognitive Function after 12 Weeks and 28 Weeks | Baseline, 12 Weeks, 28 Weeks and Up to 5 Years Post-Treatment

SECONDARY OUTCOMES:
Change from Baseline in Symptom load after 12 Weeks and 28 Weeks | Baseline, 12 Weeks, 28 Weeks and Up to 5 Years Post-Treatment
Change from Baseline in Peak oxygen uptake after 12 Weeks and 28 Weeks | Baseline, 12 Weeks, 28 Weeks and Up to 5 Years Post-Treatment
Change from Baseline in Metabolic Indices after 12 Weeks and 28 Weeks | Baseline, 12 Weeks, 28 Weeks and Up to 5 Years Post-Treatment

CONTACTS AND LOCATIONS:
Overall Officials: John A Engh, MD, PhD, Principal Investigator — Division of Mental Health & Addiction, Vestfold Hospital Trust, Tønsberg, Norway

REFERENCES:
- [Derived] Bang-Kittilsen G, Engh JA, Holst R, Holmen TL, Bigseth TT, Andersen E, Mordal J, Egeland J. High-intensity interval training may reduce depressive symptoms in individuals with schizophrenia, putatively through improved VO2max: A randomized controlled trial. Front Psychiatry. 2022 Aug 4;13:921689. doi: 10.3389/fpsyt.2022.921689. eCollection 2022. PMID 36003983
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Bang-Kittilsen G, Egeland J, Holmen TL, Bigseth TT, Andersen E, Mordal J, Ulleberg P, Engh JA. High-intensity interval training and active video gaming improve neurocognition in schizophrenia: a randomized controlled trial. Eur Arch Psychiatry Clin Neurosci. 2021 Mar;271(2):339-353. doi: 10.1007/s00406-020-01200-4. Epub 2020 Nov 6. PMID 33156372
- [Derived] Andersen E, Bang-Kittilsen G, Bigseth TT, Egeland J, Holmen TL, Martinsen EW, Stensrud T, Engh JA. Effect of high-intensity interval training on cardiorespiratory fitness, physical activity and body composition in people with schizophrenia: a randomized controlled trial. BMC Psychiatry. 2020 Aug 27;20(1):425. doi: 10.1186/s12888-020-02827-2. PMID 32854688
- [Derived] Holmen TL, Egeland J, Andersen E, Mordal J, Andreassen OA, Ueland T, Bigseth TT, Bang-Kittilsen G, Engh JA. The Association Between Cardiorespiratory Fitness and Cognition Appears Neither Related to Current Physical Activity Nor Mediated by Brain-Derived Neurotrophic Factor in a Sample of Outpatients With Schizophrenia. Front Psychiatry. 2019 Oct 25;10:785. doi: 10.3389/fpsyt.2019.00785. eCollection 2019. PMID 31708824
- [Derived] Holmen TL, Engh JA, Andersen E, Andreassen OA, Martinsen EW, Bigseth TT, Bang-Kittilsen G, Egeland J. Cardio-respiratory fitness is associated with a verbal factor across cognitive domains in schizophrenia. Schizophr Res. 2019 Apr;206:157-162. doi: 10.1016/j.schres.2018.11.033. Epub 2018 Dec 7. PMID 30528313
- [Derived] Holmen TL, Egeland J, Andersen E, Bigseth TT, Engh JA. The association between cardio-respiratory fitness and cognition in schizophrenia. Schizophr Res. 2018 Mar;193:418-422. doi: 10.1016/j.schres.2017.07.015. Epub 2017 Jul 11. PMID 28709774
- [Derived] Engh JA, Andersen E, Holmen TL, Martinsen EW, Mordal J, Morken G, Egeland J. Effects of high-intensity aerobic exercise on psychotic symptoms and neurocognition in outpatients with schizophrenia: study protocol for a randomized controlled trial. Trials. 2015 Dec 8;16:557. doi: 10.1186/s13063-015-1094-2. PMID 26646670